CLINICAL TRIAL: NCT00993486
Title: Phase I, Dose-ranging, Open-label, Study of a Single Administration of T-cells Add-back Depleted of Host Alloreactive Cells Using Theralux™ Therapy, Following Haploidentical Peripheral Blood Stem Cell Transplantation Submitted to CD34+ Cell Selection, in Patients With Severe Hematologic Malignancies
Brief Title: Dose-ranging Study of a Single Administration of T-cell Add-back Depleted of Host Alloreactive Cells in Patients Undergoing a Peripheral Blood Stem Cell Transplant From a Related, Haploidentical Donor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR-GVH-001
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Hematologic Diseases; Hematologic Malignancies
Keywords: Haploidentical stem cell transplantation; Graft-versus-host disease; Immune reconstitution; Alloreactive T-cells; Photodepletion; TH9402; Transplant related mortality; Hematologic malignancy
MeSH Terms: conditions — Hematologic Diseases; Hematologic Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- L1 (dose 1.0x10E4 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L2 (dose 5.0x10E4 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L3 (dose 1.3x10E5 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L4 (dose 3.2x10E5 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L5 (dose 7.9x10E5 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L6 (dose 2.0x10E6 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)
- L7 (dose 5.0x10E6 T-cells/kg) (Experimental)
  Interventions: Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR)

INTERVENTIONS:
Biological: Donor lymphocyte preparation depleted of functional host alloreactive T-cells (ATIR) — Single intravenous infusion

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose and evaluate the safety of the administration of donor lymphocytes depleted of alloreactive T-cells following a stem cell transplant from a related, haploidentical donor, in patients with severe hematologic malignancies.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation is the treatment of choice for many patients with leukemia and other hematologic malignancies. However, a major limitation of this therapy is that for a significant number of patients no fully HLA-matched donor can be found. The application of partially HLA-matched (haploidentical) family donors, who are virtually always available, has some complications. If there is no T-cell add-back it increases the risk for life-threatening infections and disease relapse, while in case of T-cell add-back the risk of graft-versus-host disease is raised.

Kiadis Pharma has developed a method to selectively deplete host alloreactive T-cells through photodynamic therapy, using TH9402 ex vivo. The donor lymphocyte preparation depleted of functional alloreactive T-cells (ATIR) are administered to the patient 4-6 weeks after the stem cell transplant. This method enables early immune reconstitution while preventing graft-versus-host disease.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following hematologic malignancies: very high risk leukemia, acute leukemia, chronic myeloid leukemia (CML), lymphoma, multiple myeloma (MM), myelodysplastic syndrome (MDS)
* Incompatibility at two to three loci (HLA-A, B and/or DR) or a single DR locus of the unshared haplotype between the donor and recipient
* Life expectancy of at least 3 months
* Satisfactory performance status (ECOG ≤ 2);

Exclusion Criteria:

* Possibility of performing an allogeneic transplant with an HLA (human leukocyte antigen) matched sibling donor
* Availability of an 6/6 HLA-A, B and DRB1 matched unrelated donor within 2-3 months;
* Pregnancy
* Viral hepatitis (B or C)
* Active serious infectious process
* HIV positivity;
* Systemic dysfunction (cardiac, pulmonary, hepatic and renal) contra-indicating allogeneic stem cell transplantation
* Prior allogeneic transplantation
* Prior autologous transplantation within twelve months of baseline visit
* Any abnormal condition or laboratory result that is considered by the principal investigator capable of altering patient condition or study outcome
* Active central nervous system (CNS) disease at baseline
* Participation in a trial with an investigational agent within 30 days prior to entry in the study
* Malignant cells in circulating peripheral blood (> 25%)
* Other active malignant disease that would severely limit life expectancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2005-01; Primary Completion 2008-10 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity, defined as acute graft-versus-host disease grade III or IV | Within 30 days after ATIR infusion

SECONDARY OUTCOMES:
Immune reconstitution | Until 60 months after ATIR infusion
Rate of disease relapse | Until 60 months after ATIR infusion
Occurrence and severity of graft-versus-host disease | Until 60 months after ATIR infusion
Occurrence of adverse drug reactions | Until 18 months after ATIR infusion
Incidence and severity of infections | Until 18 months after ATIR infusion

CONTACTS AND LOCATIONS:
Overall Officials: Denis-Claude Roy, MD, Principal Investigator — Maisonneuve-Rosemont Hospital, Montréal, Canada
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Roy DC, Lachance S, Cohen S, Delisle JS, Kiss T, Sauvageau G, Busque L, Ahmad I, Bernard L, Bambace N, Boumedine RS, Guertin MC, Rezvani K, Mielke S, Perreault C, Roy J. Allodepleted T-cell immunotherapy after haploidentical haematopoietic stem cell transplantation without severe acute graft-versus-host disease (GVHD) in the absence of GVHD prophylaxis. Br J Haematol. 2019 Sep;186(5):754-766. doi: 10.1111/bjh.15970. Epub 2019 May 28. PMID 31135970